CLINICAL TRIAL: NCT04828070
Title: The Heart Outcomes in Pregnancy Expectations (H.O.P.E) Registry Pilot
Brief Title: The Heart Outcomes in Pregnancy Expectations (H.O.P.E) Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HOPE Pilot Registry
Record Dates: First submitted 2020-12-02; First posted 2021-04-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Related; Cardiac Disease
Keywords: Cardio-obstetrics; HOPE Registry; Cardiac disease in pregnancy; Heart disease in pregnancy; March of Dimes
MeSH Terms: conditions — Heart Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry participant: Prospective collection of clinical information, completion of anxiety/depression, microaggressions, and quality of life questionnaires
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — all participants followed for clinical data for one year, vital status check at 5 years

SUMMARY:
Prospective US registry of pregnant women with cardiac disease to address the substantial gaps in knowledge surrounding these patients, in order to improve future care.

DETAILED DESCRIPTION:
The maternal mortality rate in the United States continues to climb, with cardiovascular disease as the leading cause for death in and around pregnancy. The racial disparities in the United States are also concerning as African American women have a 4-fold higher risk as compared to their Caucasian, Asian, or Hispanic counterparts. A Review To Action report, a collaboration of nine states' maternal mortality review committees, published in July 2018 determined that 63% of these deaths were preventable. Most deaths were related to clinical, facility and system factors, including missed or delayed diagnosis, inefficient response to obstetrical emergencies and poor communication and coordination between team members. Understanding these trends on a national level is imperative if any notable change is to be made. This requires filling the knowledge gaps that currently exist, which can be accomplished by a national registry.

Marked improvements in treating congenital heart disease have led to more women with repaired congenital cardiac malformations reaching reproductive age and desiring fertility. Beyond the growth in the prevalence of congenital heart disease, acquired cardiac disease-peripartum cardiomyopathy, ischemic heart disease, aortic dissection- are increasing and are associated with the highest risk of maternal mortality. This is particularly notable in the United States as compared to other countries where the rates of obesity and metabolic disorders approach one-third of the adult population. Adding to the complexity of the American demographics is the growing birthrate in women over 35 years of age. These trends mandate a reconceptualization of maternity care to recognize the changing demographics of pregnancy in the United States and how the growing prevalence of cardiac disease complicates care.

Other countries, particularly in Europe, have begun to investigate these issues, and as a result, their maternal mortality rates are far better than the US. Part of the European decline can be attributed to their robust prospective databases that assess pregnancy throughout the antepartum and postpartum time frame. It is becoming the dominant source of data in the medical literature describing the outcomes of patients with cardiac disease in pregnancy, yet there is no such equivalent in the United States. Investigators have yet to define the risks of pregnancy on both congenital and acquired disease states, a critical knowledge gap that could be answered with a prospective, observational registry of women with heart disease. The investigators propose to lead a prospective US registry of pregnant women with cardiac disease to address the substantial gaps in knowledge surrounding the baseline, clinical characteristics, and long-term maternal-fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Pregnant at any point in gestation (with singleton or multiple gestation)
* History of congenital and/or acquired heart disease defined as the following:

  * valvular, congenital, ischemic heart disease or cardiomyopathy,
  * clinically significant maternal arrhythmias in women,
  * current or previous history of peripartum cardiomyopathy,
  * supraventricular tachycardia,
  * placement of either a pacemaker or electrical assist device,
  * aortopathies (Marfan syndrome, Loey's Deitz, Ehlers Danlos [vascular subtype],
  * pre-pregnancy diagnosis of pulmonary hypertension
* English- or Spanish-speaking

Exclusion Criteria:

* Unable to provide written informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive outcome: Outcomes | 5 years
  Assess the maternal, neonatal and fetal outcomes of pregnancies affected by maternal cardiac disease
Descriptive outcome: morbidity and mortality | 5 years
  Assess the maternal, fetal and neonatal morbidity and mortality associated with a pregnancy that is complicated by both congenital and acquired heart disease (see inclusion criteria for these definitions) through 5 years postpartum
Descriptive outcome: quality of life parameters | 1 year
  Assess quality of life parameters during both gestation and the postpartum period in women with heart disease during pregnancy
Descriptive outcome: racial differences in maternal-fetal outcomes | 5 years
  Describe racial differences in maternal - fetal outcomes
Descriptive outcome: outcomes and care pattern changes as a result of the COVID pandemic | 5 years
  Assess the outcomes and care pattern changes as a result of the COVID pandemic for women with heart disease in pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Anna Grodzinsky, MD, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Pregnancy Mortality Surveillance System 2014. http://www.cdc.gov/reproductivehealth/maternalinfanthealth/pmss.htm
- [Background] www.Americanhealthrankings.org/explore/health-of-women-and-children/meaure/maternal_mortality/state/MO
- [Background] Blecker S, Paul M, Taksler G, Ogedegbe G, Katz S. Heart failure-associated hospitalizations in the United States. J Am Coll Cardiol. 2013 Mar 26;61(12):1259-67. doi: 10.1016/j.jacc.2012.12.038. PMID 23500328
- [Background] Siu SC, Sermer M, Colman JM, Alvarez AN, Mercier LA, Morton BC, Kells CM, Bergin ML, Kiess MC, Marcotte F, Taylor DA, Gordon EP, Spears JC, Tam JW, Amankwah KS, Smallhorn JF, Farine D, Sorensen S; Cardiac Disease in Pregnancy (CARPREG) Investigators. Prospective multicenter study of pregnancy outcomes in women with heart disease. Circulation. 2001 Jul 31;104(5):515-21. doi: 10.1161/hc3001.093437. PMID 11479246
- [Background] James AH, Jamison MG, Biswas MS, Brancazio LR, Swamy GK, Myers ER. Acute myocardial infarction in pregnancy: a United States population-based study. Circulation. 2006 Mar 28;113(12):1564-71. doi: 10.1161/CIRCULATIONAHA.105.576751. Epub 2006 Mar 13. PMID 16534011
- [Background] Khairy P, Ouyang DW, Fernandes SM, Lee-Parritz A, Economy KE, Landzberg MJ. Pregnancy outcomes in women with congenital heart disease. Circulation. 2006 Jan 31;113(4):517-24. doi: 10.1161/CIRCULATIONAHA.105.589655. PMID 16449731
- [Background] Drenthen W, Boersma E, Balci A, Moons P, Roos-Hesselink JW, Mulder BJ, Vliegen HW, van Dijk AP, Voors AA, Yap SC, van Veldhuisen DJ, Pieper PG; ZAHARA Investigators. Predictors of pregnancy complications in women with congenital heart disease. Eur Heart J. 2010 Sep;31(17):2124-32. doi: 10.1093/eurheartj/ehq200. Epub 2010 Jun 28. PMID 20584777
- [Background] Ouyang DW, Khairy P, Fernandes SM, Landzberg MJ, Economy KE. Obstetric outcomes in pregnant women with congenital heart disease. Int J Cardiol. 2010 Oct 8;144(2):195-9. doi: 10.1016/j.ijcard.2009.04.006. Epub 2009 May 2. PMID 19411123
- [Background] Liese KL, Mogos M, Abboud S, Decocker K, Koch AR, Geller SE. Racial and Ethnic Disparities in Severe Maternal Morbidity in the United States. J Racial Ethn Health Disparities. 2019 Aug;6(4):790-798. doi: 10.1007/s40615-019-00577-w. Epub 2019 Mar 15. PMID 30877505
- [Background] Daymude AEC, Catalano A, Goodman D. Checking the pregnancy checkbox: Evaluation of a four-state quality assurance pilot. Birth. 2019 Dec;46(4):648-655. doi: 10.1111/birt.12425. Epub 2019 Mar 14. PMID 30873658
- [Background] Lu MC. Reducing Maternal Mortality in the United States. JAMA. 2018 Sep 25;320(12):1237-1238. doi: 10.1001/jama.2018.11652. No abstract available. PMID 30208484
- [Background] Wolfe DS, Hameed AB, Taub CC, Zaidi AN, Bortnick AE. Addressing maternal mortality: the pregnant cardiac patient. Am J Obstet Gynecol. 2019 Feb;220(2):167.e1-167.e8. doi: 10.1016/j.ajog.2018.09.035. Epub 2018 Sep 29. PMID 30278179